CLINICAL TRIAL: NCT07199842
Title: The Effects of Dynamic Neuromuscular Stabilization Exercises in Addition to Conventional Treatment on Functional Capacity, Core Stabilization Muscle Strength, and Balance in Female Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Safiye Esin (Other)
Responsible Party: Sponsor-Investigator, Safiye Esin, Fzt.Safiye Esin, Istanbul Aydın University
Organization: Istanbul Aydın University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 28/25
Record Dates: First submitted 2025-08-13; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain, Mechanical, Biofeedback, Pain, Chronic; Low Back Pain
Keywords: Low back pain,; dynamic neuromuscular stabilization; exercise
MeSH Terms: conditions — Low Back Pain; Pain; Bronchiolitis Obliterans Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group-DNS (Experimental): DNS
  Interventions: Other: Dynamic Neuromuscular Stabilization Exercises in Addition to Conventional Treatment
- control group-Placebo (No Intervention): Placebo

INTERVENTIONS:
Other: Dynamic Neuromuscular Stabilization Exercises in Addition to Conventional Treatment — Dynamic Neuromuscular Stabilization Exercises in Addition to Conventional Treatment
  Arms: study group-DNS

SUMMARY:
Low back pain, which is currently considered a public health problem, is commonly encountered. A significant proportion of low back pain cases is of mechanical origin. "Lumbar discopathy" is a general term used to describe conditions such as Lumbar Discopathy, Lumbar Disc Herniation, Lumbosacral Radiculopathy, and internal disc injury. There are various treatment approaches available for the management of lumbar discopathy in individuals presenting with low back pain. The therapeutic effectiveness of conventional exercise in alleviating low back pain has been well-documented in the literature, and research continues on the impact of different types of exercise on low back pain. One such approach is Dynamic Neuromuscular Stabilization (DNS), which aims to restore the integrated spinal stabilization system through specific functional exercises based on the developmental kinesiological positions of a healthy infant. The DNS perspective holds that each developmental position represents an exercise position. With repetition, these exercises promote the formation of an automatic pattern of central control that becomes a fundamental component of daily movements and skills. The aim of this study is to investigate the effects of conventional physiotherapy protocols and DNS exercises applied in addition to these protocols on functional capacity, the force-generating ability of core stabilization muscles, static and dynamic balance, low back pain and lumbar functionality, and quality of life in female patients diagnosed with Lumbar Disc Herniation and experiencing chronic pain. In this study, the control group received a conventional physiotherapy program for 8 weeks, 4 days per week. The intervention group received the same conventional program plus Dynamic Neuromuscular Stabilization exercises. Outcome measures included the 6-Minute Walk Test (6MWT), core muscle strength assessment, Flamingo Balance Test, Star Excursion Balance Test (SEBT), Numeric Pain Rating Scale (NPRS), Oswestry Disability Index (ODI), and the International Physical Activity Questionnaire (IPAQ), all of which were administered before and after the treatment. As a result, statistically significant differences were observed in both the control and intervention groups when comparing pre- and post-treatment values in the NPRS, 6MWT, ODI, IPAQ, SEBT, Flamingo Balance Test, and core strength as measured by a pressure biofeedback unit. Furthermore, statistically significant differences in NPRS, ODI, and pressure biofeedback results were found in favor of the intervention group when comparing between groups. Keywords: Low back pain, DNS, Developmental Kinesiology

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 and 65 years,
* Who volunteered to participate in the study,
* Had been diagnosed with lumbar disc herniation (LDH),
* Reported a pain intensity of at least 3 on the 0-10 cm Numeric Pain Rating Scale,
* And had no specific findings such as radiculopathy or leg pain originating from LDH

Exclusion Criteria:

* Patients with a history of spinal surgery,
* Serious spinal pathologies and neurological deficits with medical contraindications to active exercise,
* A diagnosis of cancer or cooperation problems

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
6 minutes walk test | 8 weeks

SECONDARY OUTCOMES:
core muscle strength assessment, | 8 weeks
  core stabilization force measurement
Flamingo Balance Test | 8 weeks
  balance test- static
Star Excursion Balance Test (SEBT) | 8 weeks
  balance test- dynamic
Numeric Pain Rating Scale (NPRS) | 8 weeks
  pain scale
Oswestry Disability Index (ODI) | 8 weeks
  Low back disability questionnaire
International Physical Activity Questionnaire (IPAQ) | 8 weeks
  Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: gözde başbuğ, Dr. Öğr. Üyesi, Study Director — Istanbul Aydın University
Locations (1):
- İstanbul Aydın University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT07199842/Prot_000.pdf